CLINICAL TRIAL: NCT05529576
Title: Multi-factor Model Constraction for Early Warning and Diagnosis of Major Depressive Disorder
Brief Title: Multi-factor Model Constraction for Early Warning and Diagnosis of MDD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Qingdao Mental Health Center (Unknown); Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220822
Record Dates: First submitted 2022-09-01; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; Omega-3 Fatty Acids
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Major depressive disorder (Experimental): Outpatients in main-center and sub-centers; meet the DSM-IV diagnosis of Major Depressive Disorder (mental examination was conducted by at least two professional doctors); available relevant HIS system biochemical data; haven't been treated with physical therapy; age between 18-65 years old; gender is not limited.
  Interventions: Drug: Omega 3 fatty acid
- Bipolar disorder (Active Comparator): Outpatients in main-center and sub-centers; meet the DSM-IV diagnosis of Bipolar disorder (mental examination was conducted by at least two professional doctors); available relevant HIS system biochemical data; haven't been treated with physical therapy; age between 18-65 years old; gender is not limited
  Interventions: Drug: Omega 3 fatty acid
- Healthy controls (No Intervention): Healthy controls in main-center and sub-centers; no history of psychiatric disease; age between 18-65 years old; gender is not limited.

INTERVENTIONS:
Drug: Omega 3 fatty acid — Omega-3 fatty acids complementation according to the patient's CRP level
  Other Names: Ω-3 fatty acids
  Arms: Bipolar disorder; Major depressive disorder

SUMMARY:
Current research on the pathogenesis of depression shows that imbalanced inflammatory factors are closely related to Major Depressive Disorder(MDD). As reported, physical exercise, Ω-3 fatty acids, and sulforaphane can be complementary therapies for moderate-to-severe depression. In addition, imaging studies have found changes in the structure and functional connectivity of the brain. Therefore, this study intends to collect clinical and biological information from patients with depression and healthy controls to establish a multi-factor model for early warning and diagnosis of major depressive disorder

DETAILED DESCRIPTION:
The immune imbalance has been reported in patients with unipolar and bipolar depression. There is no unified conclusion in the field and severity of the immune imbalance, and the cause of cognitive impairment is unknown, which may be related to many factors. Omega-3 fatty acids are immune modulators that possess antidepressant effects.

This study includes three steps.

1. We will enroll bipolar and major depressive disorder patients who are in a depressive episode and enroll healthy controls. All subjects will be assessed at baseline
2. We will give omega-fatty acid treatment based on immune indicators
3. The follow-up will last for one year with five sessions.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients in main-center and sub-centers
* Age between 18-65 years old
* Meet the DSM-IV diagnosis of depressive episode
* HAMD-17 score>17 at baseline
* No antidepressant treatment within 6 weeks prior to enrollment
* Adequate cognition level to complete the tests necessary for the study
* Willing to sign the informed consent form

Exclusion Criteria:

* Have any contraindications to Ω-3 fatty acids
* Severe physical disease
* Diagnosed with schizophrenia, or other mental illness spectra
* Have received physical therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms assessed by HAMD-17 | up to 12 months
  Depressive symptoms are the primary outcome, and we will use HAMD-17 to examine depressive symptoms.
  Respones: a reduction of 50% or more in baseline scores.Remission:HAMD⩽7.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chen, M.D.,Ph.D, Principal Investigator — Shanghai Mental Health Center(SMHC)
Locations (1):
- Shanghai Mental Health Center IRB, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No